CLINICAL TRIAL: NCT01060007
Title: A Phase II Evaluation of Five Fractions of Radiotherapy Followed by Full Dose FOLFOX Chemotherapy as Preoperative Treatment for Rectal Cancer
Brief Title: Five Fractions of Radiotherapy Followed by Full Dose FOLFOX Chemotherapy as Preoperative Treatment for Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0696 / 201106272
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant radiation followed by FOLFOX (Experimental): Radiation - 20 Gy in 5 fractions to regional nodes. 25 Gy in the same 5 fractions to macroscopic disease. This is given over 1 week.
  FOLFOX Chemotherapy - after two weeks rest - oxaliplatin 85 mg/m2 and leucovorin 400 mg/m2 IV/2 hours followed sequentially by 5FU 400 mg/m2 IV push and 5FU 2400 mg/m2 over 46 hour CIVI. Repeat ever other week for a total of 4 courses (this equals 6 weeks).
  If 5-FU is unavailable -- oral capecitabine can be given as 1000 mg/m2 BID on days 1-7 every 14 days.
  Interventions: Radiation: External beam radiation; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-FU; Drug: Capecitabine

INTERVENTIONS:
Radiation: External beam radiation
Drug: Oxaliplatin
  Other Names: Eloxatin
Drug: Leucovorin
Drug: 5-FU
  Other Names: Fluorouracil; Efudex
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
To determine if short course radiotherapy followed by chemotherapy can maintain morbidity at or below levels reported with concurrent 5FU, oxaliplatin, and radiotherapy, while maintaining response rates comparable to what would be expected with radiotherapy and concurrent chemotherapy.

DETAILED DESCRIPTION:
Our principal objectives in this trial will be to determine if short course radiotherapy followed by chemotherapy can maintain morbidity at or below levels reported with concurrent 5FU (oral capecitabine if 5FU is unavailable), oxaliplatin, and radiotherapy, while maintaining response rates comparable to what would be expected with radiotherapy and concurrent chemotherapy. If we can establish a T stage downstaging rate that is significantly better than 50% and if acute tolerance is acceptable, then we would consider this study as having provided sufficient pilot data to support including this approach as an arm in a multi-institution phase III trial. The long-term goal is improved overall control of disease by delivering better chemotherapy earlier.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the rectum
* Patient evaluated by surgeon and found to be a potential surgical candidate. Since the primary objectives are response to chemoradiation and acute toxicity, lesions which are initially unresectable are eligible-provided the surgeon feels that, if there is sufficient response, surgery could become feasible.
* Clinical evidence of T3 or T4 disease. This can be by imaging studies (see or by physical findings (tethering on palpation for T3 lesions or invasion of a neighboring organ for T4 lesions)
* Karnofsky Performance Status at >60
* Laboratory criteria:
* Absolute neutrophil count >= 1.5 K
* Platelets >= 100 K
* Total Bilirubin <= 2.0;
* SGOT and Alkaline Phosphatase <= 2 x upper limit of normal
* Creatinine < 2.0
* Hemoglobin >= 8.0
* Informed consent signed
* Tumor measurable in at least one dimension. This may be, e.g. length and/or width measured endoscopically or on digital rectal examination, and maximum rectal wall thickness determined by imaging studies.
* Estimated longevity at least 12 months
* Patients with distant metastatic disease will be eligible if they satisfy all other conditions

Exclusion Criteria:

* Pregnant women, children < 18 years, or patients unable to give informed consent
* Patients with a past history of pelvic radiotherapy.
* Patients with any other malignancy within the past 5 years except: skin cancer or in-situ cervical cancer
* Patients with known allergy/intolerance to 5FU, Leucovorin, Oxaliplatin, Capecitabine
* Prior chemotherapy for colorectal cancer.
* Grade >= 2 peripheral neuropathy
* Any condition which, in the opinion of the treating medical oncologist, renders the patient unfit for 5FU (oral capecitabine if 5FU is unavailable), Leucovorin, Oxaliplatin chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-11; Primary Completion 2013-04 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parag Parikh, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 11/10/2009 and closed to participant enrollment on 04/18/2012.
Period: Overall Study
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Started | 80
Completed | 76
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Inevaluable for response at surgery | 3

BASELINE CHARACTERISTICS:
Groups:
- Neoadjuvant Radiation Followed by FOLFOX: Radiation - 20 Gy in 5 fractions to regional nodes. 25 Gy in the same 5 fractions to macroscopic disease. This is given over 1 week.
  FOLFOX Chemotherapy - after two weeks rest - oxaliplatin 85 mg/m2 and leucovorin 400 mg/m2 IV/2 hours followed sequentially by 5FU 400 mg/m2 IV push and 5FU 2400 mg/m2 over 46 hour CIVI. Repeat every other week for a total of 4 courses (this equals 6 weeks).
  If 5-FU is unavailable -- oral capecitabine can be given as 1000 mg/m2 BID on days 1-7 every 14 days.
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 54
Region of Enrollment [Number; unit: participants]
  United States | 76
Clinical T stage [Number; unit: participants] — * T3: Tumor invades through the muscularis propria into pericolorectal tissues
  * T4a: Tumor penetrates to the surface of the visceral peritoneum
  * T4b: Tumor directly invades or is adherent to other organs or structures
  participants
    cT3 | 69
    cT4 | 7
Clinical N stage [Number; unit: participants] — * N0: No regional lymph node metastasis.
  * N+: Metastases in 1 or greater lymph node(s)
  participants
    cN0 | 17
    cN+ | 59
Clinical M stage [Number; unit: participants] — * M0: No distant metastasis.
  * M1: Distant metastasis.
  participants
    cM0 | 69
    cM1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Rate of T Stage Downstaging
Description: T stage downstaging is defined as clinical pretreatment American Joint Committee on Cancer T stage (cT) being greater than pathologic T stage at surgery (ypT).
Time Frame: Mean number of weeks before surgery 17.3 (SD +/- 2.9 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Number analyzed (Participants) | 76
percentage of participants | 71

2. Primary Outcome: Preoperative Gastrointestinal Morbidity
Description: As measured by participants who experience grade 3 or higher gastrointestinal morbidity
Time Frame: Mean number of weeks before surgery 17.3 (SD +/- 2.9 weeks)
Population: One patient was inevaluable for primary objectives because patient withdrew consent after completing radiation therapy, refused chemotherapy, and underwent a lesion resection 7 weeks after radiation therapy.
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Number analyzed (Participants) | 79
participants | 7

3. Secondary Outcome: Incidence of Any Late Grade 3 or Higher Morbidity
Time Frame: Preoperative (mean time from start of radiation to surgery 17.3 weeks (SD +/- 2.9 weeks)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Number analyzed (Participants) | 79
participants
  Non-hematologic toxicities | 16
  Hematologic toxicities | 21

4. Secondary Outcome: Incidence of Post Chemoradiotherapy Grade 3 or Higher Morbidity
Time Frame: 1 year (completion of all treatment)
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Number analyzed (Participants) | 76
participants | 21

5. Secondary Outcome: Local Control
Description: * Kaplan-Meier projections
  * Local control = control of primary tumor
Time Frame: 30 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Number analyzed (Participants) | 76
percentage of participants | 95 [89 to 100]

6. Secondary Outcome: Rate of Overall Control
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Number analyzed (Participants) | 76
percentage of participants | 89

7. Secondary Outcome: Rate of Locoregional Control
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Number analyzed (Participants) | 76
percentage of participants | 96

8. Secondary Outcome: Freedom From Disease Relapse
Description: Kaplan-Meier projections.
Time Frame: 30 months
Population: These include all cMO evaluable cases only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Number analyzed (Participants) | 69
percentage of participants | 87 [76 to 98]

9. Secondary Outcome: Determine Quality of Anorectal Function
Description: Anorectal function was measured by the participant's response to the FACT-C questionnaire question "I have control of my bowels". The answers ranged from 0=not at all to 4=very much.
Time Frame: Up to 1 year
Population: Participants who had an ostomy were not included in this outcome measure. Participants who did not complete FACT-C questionnaire at a specific timepoint were not included in that timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-treatment | Pre-surgery | 1 Year Post-treatment
Number analyzed (Participants) | 72 | 59 | 31
Participants
  0 = not at all | 7 | 4 | 2
  1 = a little bit | 3 | 4 | 4
  2 = somewhat | 22 | 8 | 13
  3 = quite a bit | 14 | 21 | 7
  4 = very much | 26 | 22 | 5

ADVERSE EVENTS:
Description: Adverse events listed in the "Other" area have the word acute or late after the event name. Acute adverse events are followed from start of treatment until Day 90. Adverse events that occurred after Day 90 are referred to as late adverse events.
Arm/Group | Neoadjuvant Radiation Followed by FOLFOX
Serious Adverse Events (participants affected / at risk) | 4/79
Other Adverse Events (participants affected / at risk) | 79/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Radiation Followed by FOLFOX (N=79)
AST (Investigations) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Alkaline phosphatase (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chest pain (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Edema (axilla) (General disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Fever (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 4
Hypercholesteremia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
INR (Investigations) | 1
Infection with normal ANC (Infections and infestations) | 1
Leukopenia (Investigations) | 1
Lymphopenia (Investigations) | 3
Muscle spasm - bladder (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pain, Dysuria (Renal and urinary disorders) | 1
Platelets (Investigations) | 1
Port-A-Cath Pain (Surgical and medical procedures) | 1
Rigors/chills (General disorders) | 1
Sensory neuropathy (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Radiation Followed by FOLFOX (N=79)
ALT, SGPT (acute) (Investigations) | 34
ALT, SGPT (late) (Investigations) | 24
AST, SGOT (acute) (Investigations) | 35
AST, SGOT (late) (Investigations) | 30
Abdominal pain (acute) (Gastrointestinal disorders) | 19
Abdominal pain (late) (Gastrointestinal disorders) | 29
Alkaline phosphatase (acute) (Investigations) | 22
Alkaline phosphatase (late) (Investigations) | 33
Allergic reaction/hypersensitivity (late) (Immune system disorders) | 5
Anal incontinence (acute) (Gastrointestinal disorders) | 5
Anal incontinence (late) (Gastrointestinal disorders) | 6
Anorexia (acute) (Metabolism and nutrition disorders) | 36
Anorexia (late) (Metabolism and nutrition disorders) | 18
Back pain (acute) (Musculoskeletal and connective tissue disorders) | 15
Back pain (late) (Musculoskeletal and connective tissue disorders) | 4
Bladder pain (acute) (Renal and urinary disorders) | 11
Buttock pain (acute) (Musculoskeletal and connective tissue disorders) | 5
Chest pain (acute) (Cardiac disorders) | 4
Constipation (acute) (Gastrointestinal disorders) | 38
Constipation (late) (Gastrointestinal disorders) | 6
Cough (acute) (Respiratory, thoracic and mediastinal disorders) | 18
Cough (late) (Respiratory, thoracic and mediastinal disorders) | 5
Creatinine (acute) (Investigations) | 13
Creatinine (late) (Investigations) | 13
Dehydration (acute) (Gastrointestinal disorders) | 9
Dehydration (late) (Metabolism and nutrition disorders) | 8
Diarrhea (acute) (Gastrointestinal disorders) | 56
Diarrhea (late) (Gastrointestinal disorders) | 37
Dizziness (acute) (Nervous system disorders) | 26
Dizziness (late) (Nervous system disorders) | 8
Dry skin (acute) (Skin and subcutaneous tissue disorders) | 7
Dyspnea (acute) (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnea (late) (Respiratory, thoracic and mediastinal disorders) | 11
Edema: limb (acute) (General disorders) | 11
Edema: limb (late) (General disorders) | 7
Erectile dysfunction (late) (Reproductive system and breast disorders) | 6
Fatigue (acute) (General disorders) | 64
Fatigue (late) (General disorders) | 47
Fever (acute) (General disorders) | 6
Fever (late) (General disorders) | 6
Fistula, GI (late) (Gastrointestinal disorders) | 5
Flatulence (acute) (Gastrointestinal disorders) | 10
GI Leak (late) (Gastrointestinal disorders) | 4
Hair loss/alopecia (acute) (Skin and subcutaneous tissue disorders) | 14
Headache (acute) (Nervous system disorders) | 14
Headache (late) (Nervous system disorders) | 5
Heartburn/dyspepsia (acute) (Gastrointestinal disorders) | 23
Heartburn/dyspepsia (late) (Gastrointestinal disorders) | 4
Hemoglobin (acute) (Blood and lymphatic system disorders) | 75
Hemoglobin (late) (Blood and lymphatic system disorders) | 64
Hemorrhage, GI, Rectum (acute) (Gastrointestinal disorders) | 15
Hemorrhage, GI: melena (acute) (Gastrointestinal disorders) | 9
Hot flashes/flushes (acute) (Vascular disorders) | 5
Hyperbilirubinemia (acute) (Investigations) | 9
Hyperbilirubinemia (late) (Investigations) | 8
Hypercalcemia (late) (Metabolism and nutrition disorders) | 4
Hyperglycemia (acute) (Metabolism and nutrition disorders) | 34
Hyperglycemia (late) (Metabolism and nutrition disorders) | 24
Hyperkalemia (acute) (Metabolism and nutrition disorders) | 8
Hyperkalemia (late) (Metabolism and nutrition disorders) | 11
Hypoalbuminemia (acute) (Metabolism and nutrition disorders) | 47
Hypoalbuminemia (late) (Metabolism and nutrition disorders) | 45
Hypocalcemia (acute) (Metabolism and nutrition disorders) | 66
Hypocalcemia (late) (Metabolism and nutrition disorders) | 36
Hypoglycemia (acute) (Metabolism and nutrition disorders) | 4
Hypokalemia (acute) (Metabolism and nutrition disorders) | 24
Hypokalemia (late) (Metabolism and nutrition disorders) | 23
Hypomagnesemia (acute) (Metabolism and nutrition disorders) | 17
Hypomagnesemia (late) (Metabolism and nutrition disorders) | 15
Hyponatremia (acute) (Metabolism and nutrition disorders) | 41
Hyponatremia (late) (Metabolism and nutrition disorders) | 33
Hypophosphatemia (acute) (Metabolism and nutrition disorders) | 13
INR (acute) (Investigations) | 21
INR (late) (Investigations) | 6
Ileus, GI (acute) (Gastrointestinal disorders) | 9
Ileus, GI (late) (Gastrointestinal disorders) | 5
Infection - UTI (acute) (Infections and infestations) | 9
Infection with normal ANC or Grade 1 or 2 neutrophils (acute) (Infections and infestations) | 5
Infection with normal ANC or Grade 1/2 neutrophils: abdomen (acute) (Infections and infestations) | 6
Infection with normal ANC or Grade 1/2 neutrophils: skin (late) (Infections and infestations) | 4
Insomnia (acute) (Psychiatric disorders) | 26
Insomnia (late) (Psychiatric disorders) | 7
Jaw pain (acute) (Musculoskeletal and connective tissue disorders) | 5
Joint pain (acute) (Musculoskeletal and connective tissue disorders) | 6
Leak, GI (acute) (Gastrointestinal disorders) | 4
Leg pain (late) (Musculoskeletal and connective tissue disorders) | 4
Leukopenia (acute) (Investigations) | 59
Leukopenia (late) (Investigations) | 53
Lymphopenia (acute) (Investigations) | 71
Lymphopenia (late) (Investigations) | 59
Mood alteration - anxiety (acute) (Psychiatric disorders) | 27
Mood alteration - depression (acute) (Psychiatric disorders) | 15
Mood alteration-anxiety (late) (Psychiatric disorders) | 7
Mood alteration-depression (late) (Psychiatric disorders) | 5
Mucositis/stomatitis (clinical exam) (acute) (Gastrointestinal disorders) | 7
Mucositis/stomatitis (functional/symptomatic) (acute) (Gastrointestinal disorders) | 15
Mucositis/stomatitis (functional/symptomatic) (late) (Gastrointestinal disorders) | 8
Muscle pain (acute) (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness (late) (Musculoskeletal and connective tissue disorders) | 7
Nausea (acute) (Gastrointestinal disorders) | 51
Nausea (late) (Gastrointestinal disorders) | 45
Neuropathy-sensory (late) (Nervous system disorders) | 51
Neuropathy: sensory (acute) (Nervous system disorders) | 69
Neutrophils/granulocytes (acute) (Investigations) | 37
Neutrophils/granulocytes (late) (Investigations) | 30
Nose bleed (acute) (Respiratory, thoracic and mediastinal disorders) | 4
PTT (acute) (Investigations) | 16
Pain: Dysuria (acute) (Renal and urinary disorders) | 9
Perianal skin pain (acute) (Gastrointestinal disorders) | 7
Platelets (acute) (Investigations) | 45
Platelets (late) (Investigations) | 46
Pruritus/itching (acute) (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (acute) (Skin and subcutaneous tissue disorders) | 16
Rash/desquamation (late) (Skin and subcutaneous tissue disorders) | 4
Rash: dermatitis associated with radiation (acute) (Skin and subcutaneous tissue disorders) | 10
Rash: hand-foot skin reaction (acute) (Skin and subcutaneous tissue disorders) | 5
Rectal pain (acute) (Gastrointestinal disorders) | 27
Rigors/chills (acute) (General disorders) | 11
Rigors/chills (late) (General disorders) | 4
Small bowel NOS obstruction (late) (Gastrointestinal disorders) | 4
Sweating (acute) (General disorders) | 10
Taste alteration (acute) (Gastrointestinal disorders) | 11
Taste alteration (late) (Gastrointestinal disorders) | 6
Thrombosis/thrombus/embolism (Vascular disorders) | 4
Thrombosis/thrombus/embolism (acute) (Vascular disorders) | 4
Urgency, GI (acute) (Gastrointestinal disorders) | 5
Urinary frequency/urgency (acute) (Renal and urinary disorders) | 8
Urinary frequency/urgency (late) (Renal and urinary disorders) | 4
Urinary retention (acute) (Renal and urinary disorders) | 8
Urinary retention (late) (Renal and urinary disorders) | 6
Vomiting (acute) (Gastrointestinal disorders) | 24
Vomiting (late) (Gastrointestinal disorders) | 17
Weight loss (acute) (Gastrointestinal disorders) | 10
Weight loss (late) (Gastrointestinal disorders) | 14
Wound complication, non-infectious (acute) (Injury, poisoning and procedural complications) | 12
Wound complication, non-infectious (late) (Injury, poisoning and procedural complications) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes